CLINICAL TRIAL: NCT05998772
Title: Influence of Glucose on Metabolism and Clinical Symptoms of Patients With Parkinson's Disease
Acronym: PaGlu
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University of Kiel (Other)
Responsible Party: Principal Investigator, Eva Schaeffer, Principal Investigator, University Hospital Schleswig-Holstein
Other Study IDs: D 537/23
Record Dates: First submitted 2023-07-21; First posted 2023-08-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Nutritional and Metabolic Diseases; Sugar Intake
MeSH Terms: conditions — Parkinson Disease; Nutritional and Metabolic Diseases | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PD patients with craving for sweets
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Other: Placebo Oral Glucose Tolerance Test
- PD patients without craving for sweets
  Interventions: Diagnostic Test: Oral Glucose Tolerance Test; Other: Placebo Oral Glucose Tolerance Test

INTERVENTIONS:
Diagnostic Test: Oral Glucose Tolerance Test — Application of 82,5 g of glucose monohydrate solved in 300ml water
Other: Placebo Oral Glucose Tolerance Test — Application of 125mg sucralose solved in 300ml water

SUMMARY:
Many patients with Parkinson's Disease (PD) report an increased consumption of fast-acting sugars. This tendency to consume sweet, high-sugar foods occurs in some patients even before the onset of cardinal motor symptoms. Some recent studies have demonstrated that PD patients have an increased consumption of fast-acting carbohydrates compared to healthy controls. However, the reason for this change in eating behavior has not yet been adequately explained. It is discussed that the increased sugar intake leads to an increased dopamine release in the brain via an increase in insulin and thus to an improvement in clinical symptoms. This study investigates the influence of fast-acting carbohydrates on insulin and glucose blood levels as well as motor and non-motor symptoms in patients with PD using an oral glucose tolerance test and a placebo oral glucose tolerance test in a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease, stage Hoehn & Yahr 1.5-3
* Ability to pause antiparkinsonian medication in the morning without relevant impairment
* Capacity to give consent (determined in doubt by two independent neurologists, MOCA ≥18) and written informed consent.
* Patients are between 50 and 80 years of age, with exceptions for a maximum of 5 additional patients enrolled per group
* For stratification into patients with and without sweet craving, a 3-day dietary protocol should be completed once by the patients
* Group I: increased hunger for sweets.
* Group II: no increased hunger for sweets.

For the stratification into patients with and without increased hunger for sweets, participants are asked to answer the following questions:

1. Do you have sudden attacks of cravings for sweets?
2. Would you say that your consumption of sweet food has increased in recent years?
3. Would you describe your consumption of sugary food as increased or excessive?

If one of the questions is answered with yes, participants will be assigned to group I, if all questions are answered with no, participants will be assigned to group II.

Exclusion Criteria:

* Other significant neurological diseases primarily affecting the central nervous system (e.g., multiple sclerosis)
* Diagnosis of diabetes mellitus or prediabetes
* Use of medications that affect glucose metabolism, such as antidiabetics, glucocorticoids, ciclosporin, tacrolimus, sirolimus, beta-blockers, thiazide diuretics, beta-2 adrenoreceptor agonists, theophylline, Clozapine, olanzapine, paliperidone, quetiapine, risperidone, tricyclic antidepressants, mirtazapine, mianserin, carbamazepine, gabapentin, pregabalin, valproic acid, lithium, antiretroviral drugs, statins
* cardiac or brain pacemakers

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes Parkinson's Disease patients with and without sweet cravings. Recruitment of patients takes place in the outpatient clinic for movement disorders at the University of Kiel.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of Insulin in µU/mL | immediately before Application of oral glucose tolerance test and placebo as well as 30, 60, 90 and 120 minutes after application
  Blood value
Motor function | immediately before Application of oral glucose tolerance test and placebo as well as 30, 60 and 120 minutes after application
  assessed by Unified Parkinson's Disease Rating Scale Part III, 0-132 points, higher points indicate worse motor function
Concentration of Blood Glucose in mg/dL | immediately before Application of oral glucose tolerance test and placebo as well as 30, 60, 90 and 120 minutes after application
  Blood value

SECONDARY OUTCOMES:
Cognitive function | immediately before Application of oral glucose tolerance test and placebo as well as 60 minutes after application
  assessed by Montreal-Cognitive-Assessment-Test (MoCa), 0-30 points, higher points indicate better cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Neurology, University of Kiel, Kiel, Germany